CLINICAL TRIAL: NCT06503224
Title: An Exploratory Clinical Study of a Fourth-generation Autologous CAR-T Cell Injection (SCAR02) Targeting BCMA and CD19 for the Treatment of Refractory Autoimmune Diseases
Brief Title: An Exploratory Clinical Study of SCAR02 Targeting BCMA and CD19 for the Treatment of Refractory Autoimmune Diseases
Acronym: SCAR02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SWKCART24031101
Record Dates: First submitted 2024-07-07; First posted 2024-07-16 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Autoimmune Diseases
Keywords: rheumatoid arthritis; systemic lupus erythematosus; dry syndrome; systemic sclerosis
MeSH Terms: conditions — Autoimmune Diseases; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-BCMA and CD19 CART (Experimental): Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CART infusion. A dose of Anti-BCMA and CD19 CART will be infused on day 0.
  Interventions: Drug: Anti-BCMA and CD19 CART cells will be injected intravenously on a one-time basis.

INTERVENTIONS:
Drug: Anti-BCMA and CD19 CART cells will be injected intravenously on a one-time basis. — A single intravenous infusion of anti-BCMA and CD19 CART cells (dose-escalating infusion of 0.5-3 x10^6 CART cells/kg）.

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with refractory autoimmune diseases. This study aims to evaluate the safety and efficacy of the treatment with Anti-BCMA and CD19 CART

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form.
2. At the time of signing the informed consent form, the age of 18 years old or above, both male and female.
3. Bone marrow hematopoietic function is satisfied: white blood cell count ≥3×10^9/L; neutrophil count ≥1×10^9/L (not receiving colony-stimulating factor within 2 weeks prior to screening); hemoglobin ≥60g/L.
4. Liver function fulfillment: ALT≤3×ULN; AST≤3×ULN; TBIL≤3×ULN.
5. Renal function fulfillment: creatinine clearance CrCl ≥ 60mL/min.
6. Coagulation function meets: international standard ratio INR <1.5 times ULN, prothrombin time PT <1.5 times ULN.

Patients with rheumatoid arthritis must also meet the following enrollment criteria:

1. Diagnosis of rheumatoid arthritis according to the 2010 ACR / EULAR diagnostic criteria.
2. Fulfillment of one of the following conditions: DAS28-ESR >3.2 or CDAI >10 at 3 months after use of a standard treatment regimen prior to screening; inability to taper hormones (prednisone) to less than 7.5 mg/day; and number of swollen joints and/or number of joints with tenderness ≥3. Standard treatment regimen is defined as the stable use of any of the following (alone or in combination): corticosteroids, nonsteroidal anti-inflammatory drugs ( NSAIDs) and csDMARDs, including methotrexate, leflunomide, hydroxychloroquine, salazosulfapyridine, elamodex, tretinoin, and paeonia lactiflora total, as well as biological agents (including TNF inhibitors, non-TNF inhibitors, and JAK inhibitors).
3. Stable treatment with 1 or 2 cs DMARD(s) prior to enrollment as follows: at least 12 weeks of methotrexate and at least 4 weeks of administration at a dose of 7.5-25 mg/week; at least 4 weeks of stable hydroxychloroquine doses of ≤400 mg/d; at least 4 weeks of stable oral salicylazosulfapyridine 1 to 3 g/d; at least 4 weeks of stable oral leflunomide 10-20 mg /d.

Patients with SLE will also be required to meet the following enrollment criteria:

1. Diagnosis of SLE according to the 2019 EULAR/ACR classification criteria for SLE.
2. A history of SLE for at least 6 months prior to screening, with the disease remaining active 2 months after the use of a standard treatment regimen prior to screening. Standard treatment regimen is defined as stable use of any of the following (alone or in combination): corticosteroids, antimalarials, nonsteroidal anti-inflammatory drugs (NSAIDs), and other immunosuppressive or biologic agents, including azathioprine, mertiomaxolide, cyclophosphamide, methotrexate, leflunomide, tacrolimus, cyclosporine, belimumab, rituximab, and tetracycline.
3. BILAG-2004 assessment of the presence of at least 1 grade A or 2 grade B organ scores.
4. Positive for at least one of the following antibodies: anti-nuclear antibody, anti-ds-DNA antibody, anti-Sm antibody.
5. SLEDAI-2000 score ≥ 8 during the screening period.

Patients with dry syndrome were also required to meet the following enrollment criteria:

1. Diagnosis of dry syndrome according to the 2002 International Classification Criteria for Primary Dry Syndrome or the 2016 ACR/EULAR classification criteria.
2. Diagnosis of pSS-TP with platelet count <30 x 10^9/L.
3. History of dry syndrome for at least 6 months prior to screening and disease still active 2 months after use of conventional treatment regimen prior to screening. Definition of conventional therapy:Use of glucocorticoids (above 1 mg/Kg/d) and cyclophosphamide, and any of the following immunomodulatory drugs for more than 6 months: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, and cyclosporine, as well as biologics, such as rituximab, belimumab, and tetraciprazole.

Patients with systemic sclerosis were also required to meet the following enrollment criteria:

1. Diagnosis of systemic sclerosis according to the 2013 ACR classification criteria for systemic sclerosis.
2. Positive antinuclear antibodies at screening.
3. Presence of clear evidence of HRCT progression.
4. History of systemic sclerosis for at least 6 months prior to screening, and active disease 2 months after use of a conventional treatment regimen prior to screening. Definition of conventional therapy:Use of glucocorticoids (above 0.5 mg/Kg/d) and cyclophosphamide for more than 6 months, as well as any of the following immunomodulatory medications: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, and cyclosporine, as well as biologics, such as rituximab and belimumab.

Exclusion Criteria:

1. pre-screening presence of clinically significant CNS disease or pathological changes not caused by the disease itself, including, but not limited to: stroke, apoplexy, aneurysm, epilepsy, convulsions, aphasia, severe craniocerebral injury, dementia, Parkinson's disease, cerebellar disorders, organic brain syndromes, or insanity.
2. Those suffering from relatively serious heart diseases such as angina pectoris, myocardial infarction, heart failure and arrhythmia.
3. History of major organ transplantation or hematopoietic stem cell/bone marrow transplantation.
4. vaccination, B-cell targeted therapy within 4 weeks prior to screening.
5. History of any malignant disease.
6. Patients with end-stage renal failure.
7. Presence or suspected presence of uncontrolled fungal, bacterial, viral or other infections.
8. History of severe allergy to drugs used in clinical studies or raw materials of test drugs, such as cyclophosphamide, fludarabine, DMSO.
9. The patient is positive for HBV surface antigen, or HBV core antibody and positive for DNA by RT-PCR; positive for HCV antibody or positive for HIV antibody or positive for syphilis or positive for CMV DNA or positive for EBV DNA.
10. Females who are pregnant or breastfeeding or who plan to have a pregnancy within 2 years of return infusion of the test drug; partners of male patients who plan to become pregnant within 2 years of treatment with the test drug.
11. Evidence of active tuberculosis infection.
12. other circumstances assessed by the investigator as unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 2 years
  Total number, incidence and severity of adverse events (AEs) in patients of SCAR02 infusion. The AEs will be assessed according to the 2019 Consensus on Cytokine Release Syndrome and Immune-cell-associated Neurotoxicity published by the American Society of Transplantation and Cell Therapy (ASTCT), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and EBMT 2019 consensus.

SECONDARY OUTCOMES:
The persistence, accumulation, and migration of Anti-BCMA and CD19 CART cells | up to 2 years
  Assessing the trafficking of Anti-BCMA and CD19 CART cells in the peripheral blood at the time of each infusion as well as at each time of follow-up by Quantitative Real-time Polymerase Chain Reaction or flow cytometry. Peripheral blood will be collected prior to the initial infusion and will be set as baseline.
Erythrocyte Sedimentation Rate | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate disease activity
American College of Rheumatology (ACR) criteria 20, 50, 70 response rate | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate RA disease activity
Swollen and tender joint count | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate RA disease activity
Visual Analogue Scale | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate RA disease activity
Changes in the Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2000) from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  Range [0, 105]，higher score represents worse disease activity
Changes in the Physician Global Assessment (PGA) score from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  Range [0, 3]，higher score represents worse disease activity
Changes in the BILAG-2004 score from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  Range [0, 72]，higher score represents worse disease activity
Changes in immunological indexes from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  Serum IgA, IgG and IgM will be evaluated
Changes in level of anti-nuclear antibody (ANA) in peripheral blood from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate disease activity
Changes in level of anti-double stranded DNA (dsDNA) antibody in peripheral blood from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate disease activity
Changes in levels of complement in peripheral blood from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate SLE disease activity
Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24 | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate SLE disease activity
Changes in levels of anti-Ro/SSA antibodies in peripheral blood from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate disease activity
Changes in levels of Changes in levels of anti-Ro/SSA antibodies in peripheral blood from baseline in peripheral blood from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate disease activity
Changes in levels of Changes in levels of RF in peripheral blood from baseline in peripheral blood from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate disease activity
Changes in levels of Changes in levels of anti-topoisomerase I antibody in peripheral blood from baseline in peripheral blood from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate disease activity
Change in Health Assessment Questionnaire Disability Index (HAQ-DI) score from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  Change in Health Assessment Questionnaire Disability Index (HAQ-DI) describes the patient's self-assessed degree of disability. HAQ-DI comprises 8 categories of questions rated from 0 to 3, where 3 indicates the worst degree of disability.
Changes in levels of Changes in levels of anti-RNA polymerase III antibody in peripheral blood from baseline in peripheral blood from baseline | Day-1, 14, 21, 28 and Month2, 3, 6, 9, 12, 18, 24
  To evaluate disease activity

CONTACTS AND LOCATIONS:
Overall Officials: zhu chen, M.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China; xingbing wang, M.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- Hunan Siweikang Therapeutic Co.Ltd, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes